CLINICAL TRIAL: NCT06355765
Title: Effect of Oral Citicoline, Vitamins A, B, C and E, and Blackcurrant in Primary Open-Angle Glaucoma With OCT and Angiography
Brief Title: Citicoline & Antioxidants in Glaucoma
Status: Completed | Type: Observational
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Luca D'Andrea, Prinicipal investigator, University of Naples
Other Study IDs: CITIZ_001
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Citicoline blackcurrant: The treated group received a unique combination of oral dietary supplements, formulated in a soluble liquid sachet format for optimal absorption and convenience. This formulation included the following key components: citicoline (500 mg), vitamins A (300 μm), B group (4.415 mg), C (115 μm), and E (5 μm), and blackcurrant extract (50 mg). The participants in the treated group were instructed to take one sachet daily for 20 days each month, followed by a 10-day pause, and this therapy cycle was repeated throughout the 12-month follow-up period
  Interventions: Dietary Supplement: Citicoline blackcurrant supplement
- Placebo: The treated group received a unique combination of oral placebo. The participants in the treated group were instructed to take one sachet daily for 20 days each month, followed by a 10-day pause, and this therapy cycle was repeated throughout the 12-month follow-up period

INTERVENTIONS:
Dietary Supplement: Citicoline blackcurrant supplement — Citicoline, Vitamins A, B, C and E, and Blackcurrant
  Groups: Citicoline blackcurrant

SUMMARY:
To evaluate the long-term effects of oral citicoline, vitamins A, B, C and E, and blackcurrant therapy in patients with primary open-angle glaucoma (POAG) using optical coherence tomography (OCT), OCT angiography (OCTA) and microperimetry parameters.

DETAILED DESCRIPTION:
AIMS: To evaluate the long-term effects of oral citicoline, vitamins A, B, C and E, and blackcurrant therapy in patients with primary open-angle glaucoma (POAG) using optical coherence tomography (OCT), OCT angiography (OCTA) and microperimetry parameters.

METHODS: Fifteen patients with POAG (treated group) received one soluble liquid sachet daily for 20 days a month of a complementary dietary supplement containing in fixed combination citicoline, vitamins A, B, C, and E, and blackcurrant for 1 year. Fifteen age-matched subjects affected by POAG were given a placebo and served as a control group. The patients underwent best corrected visual acuity (BCVA), Goldmann applanation tonometry, microperimetry examination, OCT, and OCTA at the beginning of the study and then at 1, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of POAG
* aged between 18 and 75 years
* Patients with controlled intraocular pressure (IOP) below 20 mmHg, who had been on the same topical hypotensive therapy for at least 3 months
* myopia less than 5 diopters (D) were considered eligible for inclusion.

Exclusion Criteria:

* IOP levels exceeding 21 mmHg,
* hyper-sensitivity to citicoline,
* a history of optic neuritis,
* previous glaucoma or retinal surgery,
* prior cataract or refractive surgery,
* macular degeneration or other retinal disorders,
* any systemic diseases that could potentially lead to neurodegeneration (e.g., multiple sclerosis, diabetes)

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Ganglionar cells complex (GCC) | From enrollment to the end of treatment at 1 year
  evaluate the long-term effects of oral citicoline, vitamins A, B, C and E, and blackcurrant therapy in patients with primary open-angle glaucoma (POAG) on GCC using optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Evaluation of Retinal nerve fiber layer (RNFL) | From enrollment to the end of treatment at 1 year
  evaluate the long-term effects of oral citicoline, vitamins A, B, C and E, and blackcurrant therapy in patients with primary open-angle glaucoma (POAG) on RNFL using optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Luca D'Andrea, MD, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Italy